CLINICAL TRIAL: NCT06918145
Title: Clinical Study on the Safety, Efficacy, and Mechanisms of Lymphaticovenous Anastomosis (LVA) for the Treatment of Alzheimer's Disease (AD)
Brief Title: Clinical Study on Lymphaticovenous Anastomosis（LVA） for the Treatment of Alzheimer's Disease（AD）
Acronym: LVA; AD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006761-M20250166
Record Dates: First submitted 2025-03-23; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer&Amp;#39;s Disease (AD)
Keywords: Alzheimer's Disease（AD）; Lymphaticovenous Anastomosis（LVA）

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lymphaticovenous Anastomosis(LVA) for the Treatment of Alzheimer's Disease(AD) (Experimental)
  Interventions: Procedure: Lymphaticovenous Anastomosis

INTERVENTIONS:
Procedure: Lymphaticovenous Anastomosis — The basic principle of LVA surgery is to anastomose the deep cervical lymphatic vessels of the brain with adjacent small veins, effectively enabling the direct reflow of accumulated Aβ and tau proteins in the brain's lymphatic circulation into the venous system, thereby improving the symptoms of Alzheimer's Disease (AD).

SUMMARY:
The goal of this clinical trial is to explore the safety and efficacy of Lymphaticovenous Anastomosis (LVA) for the Treatment of Alzheimer's Disease (AD). The main questions it aims to answer are:

1. After LVA surgery treatment, do patients with AD show improvement in dementia, cognitive impairment, neurobehavioral symptoms?
2. What are the complications associated with LVA treatment for AD, including perioperative complications and long-term complications?
3. What is the mechanism of LVA treatment for AD patients, and what changes occur in AD-related biomarkers (Aβ42、 Aβ40、Aβ42/40、pTau217、pTau181) before and after surgery?

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Alzheimer's Disease based on biomarkers, imaging, and clinical symptoms;
2. Male or female aged 50-85 years (inclusive);
3. At least one caregiver who can live with the patient for an extended period;
4. No severe systemic diseases affecting the heart, liver, kidneys, etc.;
5. Patients who voluntarily participate in clinical recruitment, accept the LVA surgical treatment plan, and sign the informed consent form.

Exclusion Criteria:

1. Poor overall health, unable to tolerate surgery;
2. Preoperative anesthetic assessment indicates inability to tolerate general anesthesia;
3. Presence of other neurological or psychiatric disorders;
4. Severe bleeding tendency due to coagulopathy;
5. Inability to comply with treatment and follow-up;
6. Other conditions that preclude tolerance to surgery.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-02 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
The assessment of score changes after Lymphaticovenous Anastomosis(LVA) for the treatment of Alzheimer's Disease(AD) using Mini-Mental State Examination(MMSE). | From enrollment to the end of treatment at 3 days, 7 days, 1 month, 3 months, 6 months,1 year, 3 years, 5 years.
  The assessment of score changes by Mini-Mental State Examination(MMSE)

SECONDARY OUTCOMES:
The safety of Lymphaticovenous Anastomosis(LVA) for the Treatment of Alzheimer's Disease(AD) | From enrollment to the end of treatment at 3 days, 7 days, 1 month, 3 months, 6 months, 1 year, 3 years, 5 years.
  The complications associated with LVA treatment for AD, including perioperative complications and long-term complications.

OTHER OUTCOMES:
The mechanism of LVA treatment for AD patients | From enrollment to the end of treatment at 3 days, 7 days, 1 month, 3 months, 6 months, 1 year, 3 years, 5 years.
  The changes occur in AD-related biomarkers（Aβ42、 Aβ40、Aβ42/40、pTau217、pTau181） before and after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Formolo DA, Yu J, Lin K, Tsang HWH, Ou H, Kranz GS, Yau SY. Leveraging the glymphatic and meningeal lymphatic systems as therapeutic strategies in Alzheimer's disease: an updated overview of nonpharmacological therapies. Mol Neurodegener. 2023 Apr 20;18(1):26. doi: 10.1186/s13024-023-00618-3. PMID 37081555
- [Background] Harrison IF, Ismail O, Machhada A, Colgan N, Ohene Y, Nahavandi P, Ahmed Z, Fisher A, Meftah S, Murray TK, Ottersen OP, Nagelhus EA, O'Neill MJ, Wells JA, Lythgoe MF. Impaired glymphatic function and clearance of tau in an Alzheimer's disease model. Brain. 2020 Aug 1;143(8):2576-2593. doi: 10.1093/brain/awaa179. PMID 32705145
- [Background] Da Mesquita S, Louveau A, Vaccari A, Smirnov I, Cornelison RC, Kingsmore KM, Contarino C, Onengut-Gumuscu S, Farber E, Raper D, Viar KE, Powell RD, Baker W, Dabhi N, Bai R, Cao R, Hu S, Rich SS, Munson JM, Lopes MB, Overall CC, Acton ST, Kipnis J. Functional aspects of meningeal lymphatics in ageing and Alzheimer's disease. Nature. 2018 Aug;560(7717):185-191. doi: 10.1038/s41586-018-0368-8. Epub 2018 Jul 25. PMID 30046111
- [Background] Huang SY, Zhang YR, Guo Y, Du J, Ren P, Wu BS, Feng JF; Alzheimer's Disease Neuroimaging Initiative; Cheng W, Yu JT. Glymphatic system dysfunction predicts amyloid deposition, neurodegeneration, and clinical progression in Alzheimer's disease. Alzheimers Dement. 2024 May;20(5):3251-3269. doi: 10.1002/alz.13789. Epub 2024 Mar 19. PMID 38501315
- [Background] Chachaj A, Gasiorowski K, Szuba A, Sieradzki A, Leszek J. The Lymphatic System In The Brain Clearance Mechanisms - New Therapeutic Perspectives For Alzheimer's Disease. Curr Neuropharmacol. 2023;21(2):380-391. doi: 10.2174/1570159X20666220411091332. PMID 35410605
- [Background] Scheltens P, Blennow K, Breteler MM, de Strooper B, Frisoni GB, Salloway S, Van der Flier WM. Alzheimer's disease. Lancet. 2016 Jul 30;388(10043):505-17. doi: 10.1016/S0140-6736(15)01124-1. Epub 2016 Feb 24. PMID 26921134
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Background] Jia L, Du Y, Chu L, Zhang Z, Li F, Lyu D, Li Y, Li Y, Zhu M, Jiao H, Song Y, Shi Y, Zhang H, Gong M, Wei C, Tang Y, Fang B, Guo D, Wang F, Zhou A, Chu C, Zuo X, Yu Y, Yuan Q, Wang W, Li F, Shi S, Yang H, Zhou C, Liao Z, Lv Y, Li Y, Kan M, Zhao H, Wang S, Yang S, Li H, Liu Z, Wang Q, Qin W, Jia J; COAST Group. Prevalence, risk factors, and management of dementia and mild cognitive impairment in adults aged 60 years or older in China: a cross-sectional study. Lancet Public Health. 2020 Dec;5(12):e661-e671. doi: 10.1016/S2468-2667(20)30185-7. PMID 33271079